CLINICAL TRIAL: NCT01931878
Title: Investigation of Efficacy of incobotulinumtoxinA (Xeomin) in Relieving Symptoms of Restless Leg Syndrome.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1206010332
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Restless Leg Syndrome
Keywords: Restless Legs Syndrome; Leg pain; Sleep; Dysesthesias; incobotulinumtoxin
MeSH Terms: conditions — Restless Legs Syndrome; Paresthesia | interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo , saline (Placebo Comparator): The subject may be randomly assigned to receive Placebo, saline
  Interventions: Drug: Placebo
- IncobotulinumtoxinA Treatment (Active Comparator): The subjects will be randomized to received injections of active study drug, incobotulinumtoxinA (Xeomin)
  Interventions: Drug: incobotulinumtoxinA

INTERVENTIONS:
Drug: incobotulinumtoxinA — The subject may be randomly assigned to receive incobotulinum toxinA (Xeomin) , a neurotoxin Which is approved for use by the FDA for certain conditions. This study has a double blind cross over design. Cross over means that you will have two sets of injections. If the first set of injections is Xeomin, the second injections after a three month interval will be the inactive placebo. Double blind means neither the investigators nor the subject knows which one of the two (Xeomin or placebo) is received with the first or second injections.
  Other Names: Xeomin
  Arms: IncobotulinumtoxinA Treatment
Drug: Placebo — The subject may be randomly assigned to receive Placebo which is an inactive test substance which has no active ingredient. In this protocol we use sterile salt water as placebo.This study has a double blind cross over design. Cross over means that you will have two sets of injections. If the first set of injections is placebo, the second injections after a three month interval will be active study drug. Double blind means neither the investigators nor the subject knows which one of the two (Xeomin or placebo) is received with the first or second injections.
  Other Names: Sterile saline water
  Arms: Placebo , saline

SUMMARY:
The purpose of this research study is to compare the safety and effectiveness of local injections of botulinum toxin A (Xeomin®) to an inactive test substance (placebo) in a medical condition called Restless Leg Syndrome. This study has a double blind cross over design. Cross over means that you will have two sets of injections. The first set of injections can be either Xeomin or placebo. The order of injection will be reversed at the three month point following the first injection. Double blind means neither the investigators nor you know which one of the two (Xeomin or placebo) you received.

DETAILED DESCRIPTION:
Please contact the PI for details about the clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18- 80 years of age, both sexes, all races and ethnic groups.
* Diagnosis of restless legs syndrome
* Disease duration longer than 3 months
* Restless Leg Syndrom Rating Scale score of 11 or above (moderate and above)
* Subjects who are eligible to be treated with a botulinum toxin for a therapeutic reason based upon the physicians' clinical experience.
* Subjects who are able to read, speak, and understand English.

Exclusion Criteria:

* Existing significant acute medical condition (i.e. cardiovascular, endocrine, hematologic, neoplastic, infectious, or autoimmune disorders).
* Pregnancy or planned pregnancy (determined by urine pregnancy test). Women of childbearing age should use a reliable mode of contraception during the study period (abstinence, etc).
* Active breast feeding.
* Enrollment in any clinical trial (currently or within the past 3 months) in which treatments are imposed by a protocol.
* Any subject for whom botulinum toxin treatment would be contraindicated; known allergy or sensitivity to medication.
* Subjects who are younger than 18 years of age.
* Neuromuscular-junction disorders.
* Evidence of acute pathology by neuro-imaging.
* Axis I diagnosis determined by a neurologist or psychiatrist.
* Anesthetic medications within two weeks and corticosteroid injections within 4 weeks of enrollment.
* Subject has received botulinum toxin injections in the past 4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bahman Jabbari, MD, Principal Investigator — Yale University
Locations (1):
- Yale Physcian Building, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Mittal SO, Machado D, Richardson D, Dubey D, Jabbari B. Botulinum Toxin in Restless Legs Syndrome-A Randomized Double-Blind Placebo-Controlled Crossover Study. Toxins (Basel). 2018 Sep 29;10(10):401. doi: 10.3390/toxins10100401. PMID 30274305

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First, Then Incobotulinumtoxin A: Placebo: The subject may be randomly assigned to receive Placebo which is an inactive test substance which has no active ingredient. In this protocol we use sterile salt water as placebo.This study has a double blind cross over design. Cross over means that you will have two sets of injections. If the first set of injections is placebo, the second injections after a three month interval will be active study drug.
- IncobotulinumtoxinA First, Then Placebo: The subjects will be randomized to received injections of active study drug, incobotulinumtoxinA (Xeomin)
  incobotulinumtoxinA: The subject may be randomly assigned to receive incobotulinum toxinA (Xeomin) , a neurotoxin Which is approved for use by the FDA for certain conditions. This study has a double blind cross over design. Cross over means that you will have two sets of injections. If the first set of injections is Xeomin, the second injections after a three month interval will be the inactive placebo.
Period: First Intervention
Arm/Group | Placebo First, Then Incobotulinumtoxin A | IncobotulinumtoxinA First, Then Placebo
Started | 10 | 14
Completed | 9 | 14
Not Completed | 1 | 0
Period: Second Intervention (After 3 Months)
Arm/Group | Placebo First, Then Incobotulinumtoxin A | IncobotulinumtoxinA First, Then Placebo
Started | 9 | 14
Completed | 9 | 12
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Cross over study. total 24 enrolled , 21 completed. The twenty one who competed the study had both saline and incobotulinum toxin injection ( crossover).
Groups:
- All Study Participants: The subject may be randomly assigned to receive Placebo, saline
  Placebo: The subject may be randomly assigned to receive Placebo which is an inactive test substance which has no active ingredient. In this protocol we use sterile salt water as placebo.This study has a double blind cross over design. Cross over means that you will have two sets of injections. If the first set of injections is placebo, the second injections after a three month interval will be active study drug. Double blind means neither the investigators nor the subject knows which one of the two (Xeomin or placebo) is received with the first or second injections.
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.71 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Restless Leg Syndrome Rating Scale Score
Description: The Restless Legs Syndrome Rating Scale uses 10 questions, each scored 0-4, with higher scores representing more severe symptoms. Score ranges from 1-40. Scoring criteria are: Mild (score 1-10); Moderate (score 11-20); Severe (score 21-30); Very severe (score 31-40)
Time Frame: 6 weeks
Population: Total RLS scale score was compared between incoA injections and and saline group injections.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: In this protocol we use sterile salt water as placebo.This study has a double blind cross over design. Cross over means that you will have two sets of injections.
- Xeomin: incobotulinumtoxinA: The subject may be randomly assigned to receive incobotulinum toxinA (Xeomin) , a neurotoxin which is approved for use by the FDA for certain conditions. This study has a double blind cross over design.
Arm/Group | Placebo | Xeomin
Number analyzed (Participants) | 21 | 21
units on a scale | 25.19 (7.82) | 19.46 (9.41)
Statistical Analysis 1: Comparison: Placebo vs Xeomin; comparison of mean RLS Scale scores between 21 incoA and 21 saline injections; Test type: Superiority or Other; p = 0.031, t-test, 2 sided

2. Other Pre Specified Outcome: Patients With Pain on Visual Analog Scale <4
Description: The Visual Analog Scale (VAS) consists of a line which represents the level of pain in 10 cms. The subject is required to make this line to show where your pain level is on this line (for example, at the 7cm mark). A higher score is associated with a higher level of pain. Number of patients showing a pain score of <4.
Time Frame: 6 weeks
Measure: Number; unit: participants
Groups:
- Placebo: The subject may be randomly assigned to receive Placebo, saline
  Placebo: The subject may be randomly assigned to receive Placebo which is an inactive test substance which has no active ingredient. In this protocol we use sterile salt water as placebo.
- Xeomin: The subjects will be randomized to received injections of active study drug, incobotulinumtoxinA (Xeomin)
  incobotulinumtoxinA: The subject may be randomly assigned to receive incobotulinum toxinA (Xeomin) , a neurotoxin Which is approved for use by the FDA for certain conditions.
Arm/Group | Placebo | Xeomin
Number analyzed (Participants) | 21 | 21
participants | 3 | 12
Statistical Analysis 1: Comparison: Placebo vs Xeomin; Test type: Superiority or Other; p = 0.0088, Fisher Exact

3. Secondary Outcome: Number of Patients Whose Patient Global Impression of Change (PGIC) Moderately or Much Improved
Description: The PGIC is a 7 point scale that requires the clinician to assess how much the patient's pain has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as:
  No change (or condition has gotten worse) (1) Almost the same, hardly any change at all (2) A little better, but no noticeable change (3) Somewhat better, but the change has not made any real difference (4) Moderately better, and a slight but noticeable change (5) Better and a definite improvement that has made a real and worthwhile difference (6) A great deal better and a considerable improvement that has made all the difference (7)improved
  This outcome is number of patients who chose a 5 or above on the PGIC 6 weeks after treatment.
Time Frame: 6 weeks
Measure: Number; unit: participants
Groups:
- Placebo , Saline: Placebo: The subject may be randomly assigned to receive Placebo which is an inactive test substance which has no active ingredient. In this protocol we use sterile salt water as placebo.This study has a double blind cross over design.
- IncobotulinumtoxinA Treatment: incobotulinumtoxinA: The subject may be randomly assigned to receive incobotulinum toxinA (Xeomin) , a neurotoxin Which is approved for use by the FDA for certain conditions. This study has a double blind cross over design.
Arm/Group | Placebo , Saline | IncobotulinumtoxinA Treatment
Number analyzed (Participants) | 21 | 21
participants | 3 | 9
Statistical Analysis 1: Comparison: Placebo , Saline vs IncobotulinumtoxinA Treatment; Test type: Superiority or Other; p = 0.0855, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo , Saline | IncobotulinumtoxinA Treatment
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

LIMITATIONS AND CAVEATS:
Relatively small number of participants. crossover not parallel design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No